CLINICAL TRIAL: NCT01676844
Title: Oral Potassium Acid Phosphate Supplementation for Preterm Neonates; a Comparison of Oral Thin Films and Standard Oral Therapy.
Brief Title: Investigating a New Way of Giving Medicine to Newborn and Preterm Babies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Strathclyde (Other)
Responsible Party: Principal Investigator, Professor Alex Mullen, Principal Investigator, University of Strathclyde
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UEC1112/65; 2012-003625-19 (EudraCT Number)
Record Dates: First submitted 2012-08-23; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Hypophosphataemia; Osteopenia of Prematurity
Keywords: Phosphorus; Phosphate; Hypophosphataemia; Osteopenia; Prematurity
MeSH Terms: conditions — Hypophosphatemia; Bone Diseases, Metabolic; Premature Birth | interventions — Standard of Care; potassium phosphate; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral thin film therapy (Experimental): One or more oral thin films (OTFs) containing potassium acid phosphate administered to the inside cheek, tongue or palate at a dose of 0.5 mmol/kg body weight twice daily. Dosages will be rounded to the nearest 0.1 mM/kg. Where more than one OTF is required to achieve a dosage of 0.5mmol/kg, strips will be administered consecutively with time allowed between doses to allow for complete dissolving of the previous strip. Treatment will continue until the participant has received OTF therapy for 14 consecutive days.
  Interventions: Drug: Oral thin film therapy (Potassium acid phosphate oral thin films)
- Standard therapy (Active Comparator): Standard oral phosphate supplementation as per NHS Greater Glasgow and Clyde Guidelines. An oral solution containing potassium acid phosphate (1 mmol/mL) will be administered at a dosage of 0.5 mM/kg body weight twice daily. Dosages will be rounded to the nearest 0.1 mM/kg. Standard therapy will continue until the participant has received treatment for 14 consecutive days.
  Interventions: Drug: Standard therapy (Potassium acid phosphate oral solution)

INTERVENTIONS:
Drug: Oral thin film therapy (Potassium acid phosphate oral thin films) — Orally dissolving thin film. White, square oral thin film. 15 mm x 15 mm surface area. 1-2 mm film thickness. No markings.
  Place a single OTF on the tongue, inside cheek or palate and allow to dissolve.
  Other Names: Potassium acid phosphate oral thin films 0.2, 0.3 and 0.4 mM
  Arms: Oral thin film therapy
Drug: Standard therapy (Potassium acid phosphate oral solution) — Each millilitre contains approximately 136mg Monobasic Potassium Phosphate Ph.Eur. (KH2PO4) equivalent to 1mmol Potassium (39mg) and 1mmol Phosphate (31mg Phosphorus). Manufacturer: Specials Products Ltd., Surrey, UK.
  Other Names: Potassium acid phosphate 1mmol in 1ml oral solution
  Arms: Standard therapy

SUMMARY:
There is a deficit in the number of 'age-appropriate' formulations available for the delivery of medicines to children. Liquid preparations are considered the 'gold standard' for delivering medicines to children however many of these are formulated using ingredients which can be toxic to children (e.g. preservatives, alcohols), particularly to neonatal babies (< 4 weeks old) who do not possess the metabolic processes and mature organ function of older children or adults. Rapidly dissolving oral thin films (OTFs) dissolve quickly in the saliva, releasing the active ingredient(s) without the need for chewing or water, making them ideally suited to patients who find it difficult to swallow other oral dosage forms such as tablets or capsules. The aim of this study is to demonstrate that OTFs can offer a safe and effective alternative for oral administration of phosphate supplements to neonatal infants for the treatment of hypophosphataemia and osteopenia of prematurity. It is hypothesised that this treatment will be equal to standard therapy using an oral solution. Babies born before 32 weeks gestational age are routinely supplemented with oral phosphate as soon as they have been established on oral feeds in order to prevent bone disorders such as osteopenia. Babies recruited to this study will be given phosphate supplementation as per NHS Greater Glasgow and Clyde guidelines. This single-centre cross-over study will take place in the intensive care and special care baby units at the Princess Royal Maternity in Glasgow. The investigators aim to recruit 20-30 babies and will use blood phosphate levels (obtained from routine sampling only) to evaluate treatment effect. Babies will be randomised to receive either OTFs or oral solution of potassium acid phosphate for 2 weeks followed by 2 weeks of the other therapy. The investigators hypothesise that OTF treatment will be equivalent to standard oral solution.

DETAILED DESCRIPTION:
There is a lack of 'age-appropriate' formulations available for delivering medicines to children. Liquid formulations are considered the 'gold standard' for delivering medicines to children. However, many of these are formulated using ingredients which can be toxic to children, and particularly to neonates (children <4 weeks old), who do not possess the metabolic processes and mature organ function of adults. For example, many liquid formulations contain preservatives such as benzoic acid to improve the shelf-life of the product, or include solvents such as propylene glycol or ethanol to improve solubility. Many of these additional, functional ingredients can product toxic effects in children. For example, neonates are unable to metabolise benzoic acid, resulting in the accumulation of this ingredient and potentially serious neurological and respiratory effects known as 'gasping syndrome'. Additionally, the lack of suitable licensed formulations for children leads to the routine prescribing of medicines outside the terms of their product license and/or the manipulation of medicines to make them suitable for children e.g. grinding up tablets. Further manipulation of products increases the risk of inaccurate dosages being administered, and adds a risk of error where additional calculations are required. There are also concerns over compatibility when medicines are, for example, mixed with foods or drinks in an attempt to improve acceptability. Looking specifically at prescribing within neonatal intensive care, up to 90% of medicines prescribed are unlicensed or off-label i.e. used in a way not covered by the product licence. Therefore, there is a need for more age-appropriate solid formulations suitable for delivering medicines to children. By formulating the medicine in a solid dosage form, the need for excipients such as preservatives can be removed. Within the last few years, rapidly dissolving oral thin films (OTFs) have been developed as a novel solid dosage platform for drug delivery. They were first established as breath fresheners and have since progressed towards delivery of active pharmaceutical ingredients (APIs). Approximately the size of a postage stamp, OTFs dissolve quickly in the saliva, releasing the drug(s) without the need for chewing or water. They are ideally suited to patients who find it difficult to swallow other oral dosage forms such as tablets or capsules. Paediatric and elderly patients are particularly suited to this dosage design. Flavourings and sweeteners can be included in the films to mask a bitter tasting medicine if necessary. The films are discreet, easy to use and convenient. They have a history of uses in oral hygiene products and medical devices. Recent developments have seen their use in over-the-counter cough and cold remedies and anti-allergy products. In 2010, Zuplenz® became the first FDA approved prescription only medicine in an OTF formulation for the delivery of ondansetron in the treatment of chemotherapy-induced nausea and vomiting. Most recently in February 2012, Applied Pharma Research (APR) were successful in marketing a prescription only zolmitriptan based OTF product for the treatment of migraine. A basic thin film formulation can contain very few ingredients and since they are presented as a solid dosage form, they do not require the addition of preservatives. In the USA, Novartis has already marketed several thin film products under the brand Triaminic® which are aimed at children from as young as four for the treatment of coughs, colds, and allergies. In order to investigate whether OTFs are a safe alternative for drug delivery to neonates, an OTF containing potassium acid phosphate (KAP) has been formulated. KAP was chosen for this study since it is a non-toxic mineral supplement routinely given to preterm infants to improve bone health. The majority of fetal uptake of calcium and phosphorus occurs during the third trimester of pregnancy and so preterm infants are born with reduced body stores of these minerals. Hypophosphataemia (low blood phosphorus) results in increased levels of calcitriol, the active form of vitamin D, and subsequent demineralisation of bone (osteopenia). The association between low birth weight, hypercalcaemia (high blood calcium) and hypophosphataemia was first identified in the early 1980s. It was identified that active demineralisation of bone was occurring in order to maintain the blood levels of phosphate required for other cellular functions and tissue growth. Reduced bone mineral density or metabolic bone disease in very low birth weight premature infants can lead to complications such as fractures and reduced growth. Preterm infant milk formulas and human breast milk fortifiers are supplemented with phosphate, and in addition within NHS Greater Glasgow and Clyde it is routine clinical practice to provide all preterm infants born before 32 weeks' gestational age with an oral phosphate supplement.

ELIGIBILITY:
Inclusion Criteria:

* GENDER Male or female
* AGE Born < 32 completed weeks' gestational age
* CONSENT Parents/other caregivers demonstrate understanding of the study and willingness to consent to their child's participation as evidenced by voluntary written informed consent (signed and dated) obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* MEDICATIONS AND TREATMENTS Participants must have been established on oral feeds (as defined by as > 75% of predicted volume enterally for three consecutive days).

Exclusion Criteria:

* MEDICATIONS Patients prescribed concomitant medication known to interact with potassium phosphate or any of the other ingredients in the oral thin film.
* CLINICAL STUDIES

  * Previous participation in this study.
  * Subject whose participation in this study will result in a participation in more than four studies over a twelve month period.

Ages: 26 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Serum phosphate | Participants will be followed from birth until the end of the study period, approximately 6 weeks on average
  The aim of this research is to demonstrate that oral thin films (OTFs) containing potassium acid phosphate are equivalent to standard oral phosphate supplementation using an oral solution in the prevention of hypophosphataemia (low blood phosphorus). The primary outcome measure will be plasma phosphate. We will assume an equivalent therapeutic effect using OTFs if individual plasma levels for these babies are found to lie within an acceptable physiological range, and the difference between the means of the two groups (as determined by a statistical t-test) lies within 20% of the mean plasma level for the control group.

SECONDARY OUTCOMES:
Age-appropriateness | Participants will be followed from birth until the end of the study period, approximately 6 weeks on average
  Secondary objectives will be in terms of age-appropriateness and general acceptability. A lack of any observable adverse effects e.g. choking, vomiting, diarrhoea, will indicate the safety of oral thin films in this age group. Acceptability will be assessed in terms of observed discomfort/distress e.g. grimacing, crying, associated with treatment administration and will be assessed using visual analogue scales.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Mullen, Principal Investigator — University of Strathclyde
Locations (1):
- Princess Royal Maternity, Glasgow, Strathclyde, United Kingdom

REFERENCES:
- [Background] Conroy S, McIntyre J. The use of unlicensed and off-label medicines in the neonate. Semin Fetal Neonatal Med. 2005 Apr;10(2):115-22. doi: 10.1016/j.siny.2004.11.003. Epub 2005 Jan 25. PMID 15701577
- [Background] Lyon AJ, McIntosh N, Wheeler K, Brooke OG. Hypercalcaemia in extremely low birthweight infants. Arch Dis Child. 1984 Dec;59(12):1141-4. doi: 10.1136/adc.59.12.1141. PMID 6441525
- [Background] Mitchell SM, Rogers SP, Hicks PD, Hawthorne KM, Parker BR, Abrams SA. High frequencies of elevated alkaline phosphatase activity and rickets exist in extremely low birth weight infants despite current nutritional support. BMC Pediatr. 2009 Jul 29;9:47. doi: 10.1186/1471-2431-9-47. PMID 19640269
- [Background] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Background] Marks J, Srai SK, Biber J, Murer H, Unwin RJ, Debnam ES. Intestinal phosphate absorption and the effect of vitamin D: a comparison of rats with mice. Exp Physiol. 2006 May;91(3):531-7. doi: 10.1113/expphysiol.2005.032516. Epub 2006 Jan 23. PMID 16431934
- [Background] Walton J, Gray TK. Absorption of inorganic phosphate in the human small intestine. Clin Sci (Lond). 1979 May;56(5):407-12. doi: 10.1042/cs0560407. PMID 477225
- [Background] Chen TC, Castillo L, Korycka-Dahl M, DeLuca HF. Role of vitamin D metabolites in phosphate transport of rat intestine. J Nutr. 1974 Aug;104(8):1056-60. doi: 10.1093/jn/104.8.1056. No abstract available. PMID 4854171
- [Background] Uribarri J. Phosphorus homeostasis in normal health and in chronic kidney disease patients with special emphasis on dietary phosphorus intake. Semin Dial. 2007 Jul-Aug;20(4):295-301. doi: 10.1111/j.1525-139X.2007.00309.x. PMID 17635818
- [Background] Borowitz SM, Ghishan FK. Phosphate transport in human jejunal brush-border membrane vesicles. Gastroenterology. 1989 Jan;96(1):4-10. doi: 10.1016/0016-5085(89)90757-9. PMID 2909436